CLINICAL TRIAL: NCT01138254
Title: The Effect of Far Infrared (FIR) Therapy on Access Flow of Arteriovenous (AV) Fistula, Echocardiographic Parameters and Endothelial Function in Patients With End Stage Renal Disease
Brief Title: Far Infrared Therapy on AV Fistula Flow, Endothelial Function and Echocardiography in ESRD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: CHIH-CHING LIN, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V98C1-045
Record Dates: First submitted 2010-05-25; First posted 2010-06-07 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: End Stage Renal Disease
Keywords: flow,echocardiography,far infrared therapy,nitric oxide
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): ESRD patients will not receive FIR therapy in this study.
  Interventions: Other: no intervention
- Far infrared therapy (Experimental): Patients will receive far infrared therapy 40 minutes three times weekly (TIW) for 6 months.
  Interventions: Device: WSTM TY101 FIR emitter (Far infrared therapy)

INTERVENTIONS:
Device: WSTM TY101 FIR emitter (Far infrared therapy) — A WSTM TY101 FIR emitter (WS Far Infrared Medical Technology Co., Ltd., Taipei, Taiwan) will be used for FIR therapy. The electrified ceramic plates of this emitter generate electromagnetic waves with wavelengths in the range between 3 and 25 μm (a peak between 5 to 6 μm). The irradiating power density is 10 and 20 mili watt<mw>/cm2 when the top radiator is set at a distance between 30 and 20 cm above the skin surface respectively. In this study, the top radiator will be set at a height of 25 cm above the surface of bilateral lower legs and the treatment time will be set at 40 minutes three times weekly (TIW) for ESRD patients for 6 months.
  Other Names: Far infrared therapy (WSTM TY101 FIR emitter)
  Arms: Far infrared therapy
Other: no intervention — no intervention
  Other Names: no intervention by FIR therapy
  Arms: control group

SUMMARY:
Vascular access complications are the leading cause of morbidity in hemodialysis (HD) patients, and are responsible for a significant percentage of hospitalization, with annual costs approaching one billion dollars in the United States. Thrombosis is the most common cause of vascular access failure, and usually develops from stenotic lesions in the venous outflow tract. It has been reported that far infrared (FIR) therapy can improve access flow and unassisted patency of AV fistula, however, the effect of FIR on cardiac function is unknown.

The aims of this study are to evaluate (1) the change of access flow of AV fistula and the effect of AV fistula on echocardiographic parameters and (2) the effect of FIR on access flow of AVF and echocardiographic parameters and the serum levels of endothelial markers in patients with end stage renal disease (ESRD) during the first 6 months after the creation of AV fistula.

DETAILED DESCRIPTION:
For patients with end stage renal disease receiving hemodialysis (HD) treatment, a well-functioning vascular access is necessary for achieving adequate dialysis and improving the quality of life. Among several types of vascular access, the long-term technical survival is best for the native arteriovenous fistula (AVF), which accounts for more than 80% of vascular access in HD patients in Taiwan. Vascular access complications accounted for about 20% of HD patient hospitalizations in the United States with a cost of $1 billion annually (1). Malfunction of vascular access usually presents with inadequate blood flow because of stenosis or thrombosis of the venous outflow tract (2). About 80 to 85% of AV access failures arise from AV access thromboses, of which more than 80% result from AVF stenoses (3). An access flow (Qa) less than 500 ml/min was associated with an increased risk of access failure and predictive of poorer unassisted patency of native AVF (4). The pathological features of stenosis of vascular access are composed of intimal hyperplasia; proliferation of smooth muscle cells in the media with subsequent migration to intima, and excessive accumulation of extracellular matrix (5). In spite of the above findings, little information is available on how to effectively prevent the stenoses of vascular access in HD patients.

Infrared radiation is an invisible electromagnetic wave with a longer wavelength than that of the visible light. According to the difference in wavelength, infrared radiation can be divided into three categories: near-infrared radiation (0.8-1.5μm), middle-infrared radiation (1.5-5.6μm) and far-infrared (FIR) radiation (5.6-1000μm) (6). Infrared radiation transfers energy that is perceived as heat by thermo- receptors in the surrounding skin (7). The application of FIR radiation includes food preservation (8) and health promotion (9-10). Animal studies also demonstrated that FIR improves skin blood flow(11-12), leading to the use of FIR in the treatment of ischemic lesions and necrosis of skin tissue due to trauma, diabetes mellitus and peripheral arterial occlusive disease. In addition, some studies indicate that FIR therapy may improve endothelial function and reduce the frequency of some cardiovascular diseases (13-15). The thermal effect of FIR results in vasodilatation and may increase access flow of AV fistula. According to the report by Vaupel et al., the temperature can be increased up to 4°C in 10 mm depth of tissue (16). In addition, infrared therapy may allow multiple energy transfer as deep as 2-3 cm into subcutaneous tissue without irritating or overheating the skin like unfiltered heat radiation (17). The skin temperature steadily increased to a plateau around 38~39 °C during the treatment of FIR for 30 to 60 minutes as long as the distance between the ceramic plate and the skin was more than 20 cm (11). Therefore, infrared therapy can be free of the disadvantages or side effects (such as burn injury, infection, risk of access failure or prolonged bleeding from the previous venopuncture site) of some traditional methods of thermal therapy.

In addition to the thermal effect, three possible non-thermal effects of infrared therapy were reported in the literature, including (1) improving endothelial function, (2) inhibiting intimal hyperplasia, and (3) decreasing oxidative stress. FIR may improve endothelial function which is observed not only in animal studies (11,12,14) but also in one clinical study (13). Yu et al. suggest that the beneficial effect of FIR therapy on skin blood flow may be related to L-arginine/NO pathway (11). In this respect, Akasaki et al. found that repeated FIR therapy could up-regulate eNOS expression and augment angiogenesis in an apolipoprotein E-deficient mouse model of unilateral hind limb ischemia (12). Moreover, Ikeda et al. reported that 4 weeks of sauna therapy significantly increased the serum nitrate concentrations as well as the expression of mRNA and protein of eNOS in the aortas of TO-2 hamsters (14). In addition, Imamura et al. showed that two weeks of repeated sauna therapy significantly improved vascular endothelial function, resulting in an increase in flow-mediated endothelium-dependent dilatation of the brachial artery from 4% to 5.8% in patients with coronary risk factors (13).

In addition to enhancing eNOS expression, Kipshidze et al. found that nonablative infrared laser (NIL) therapy inhibited neointimal hyperplasia after PTCA in cholesterol-fed rabbits for up to 60 days (18). According to their report, the nonablative doses of NIL decreased the growth of vascular smooth muscle cells (VSMC), but it did not decrease the growth rate of endothelial cells. As the proliferation of VSMCs in the media is an important pathological finding of the vascular wall of HD patients with vascular access stenosis (5), slowing down the growth of VSMCs may reduce the frequency of access stenosis. According to the report by Masuda et al. (19), the systolic blood pressure and the increased urinary 8-epi-prostaglandin F2α levels were significantly lower in the patients receiving an FIR dry sauna for 45 minutes per day for two weeks. F2-isoprostanes, namely 8-epi-prostaglandin F2α, are chemically stable products of lipid peroxidation and the level has been suggested as a reliable marker of oxidative stress in vivo (20). These results suggest that repeated sauna therapy may reduce oxidative stress, which leads to protection against the progression and complications of atherosclerosis. Since HD patients are also exposed to heavy oxidative stress from both inward uremic status and outward HD-related technology, the application of FIR therapy may be considered as an alternative therapeutic modality for decreasing oxidative stress.

Nakhoul et al. have shown a high incidence of unexplained pulmonary hypertension (PHT) in end-stage renal disease (ESRD) patients on chronic haemodialysis (HD) therapy via arterio-venous (A-V) access [21]. Pulmonary artery pressure (PAP) was evaluated using Doppler echocardiography. Levels of ET-1 and NO metabolites in plasma were determined before and after the HD procedure and were compared between subgroups of patients with and without PHT. Out of 42 HD patients studied, 20 patients (48%) had higher PHT (PAP = 46+/-2 mmHg) while the rest had a normal PAP (29+/-1 mmHg) (P<0.0001). In comparison with HD patients without PHT, HD patients with PHT had higher cardiac output (6.0+/-1.2 vs 5.2+/-0.9 l/min, P<0.034), similar plasma ET-1 levels (1.6+/-0.7 vs. 2.4+/-0.8 fmol/ml), lower basal plasma levels of NO2 + NO3 (14.3+/-2.3 μM vs. 24.2+/-5.2μM, P<0.05), and a lower HD-induced increase of plasma NO metabolites (from 14.3+/-2.3 to 39.9+/-11.4 microM, P<0.007 vs. from 24.2+/-5.2 to 77.1+/-9.6μM, P<0.0001, respectively). Temporary closure of the A-V access by a sphygmomanometer in eight patients with PHT resulted in a transient decrease in CO (from 6.4+/-0.6 to 5.3+/- 0.5 l/min, P = 0.18) and systolic PAP (from 47.2+/-3.8 to 34.6+/-2.8 mmHg, P<0.028). In summary, their study demonstrated a high prevalence of PHT among patients with ESRD on chronic HD via a surgical A-V fistula. In view of the vasodilatory and antimitogenic properties of NO, it is possible that the attenuated basal and HD-induced NO production in patients with PHT contributes to the increased pulmonary vascular tone. Furthermore, the partial restoration of normal PAP and CO in HD patients that underwent either temporal A-V shunt closure or successful transplantation indicates that excessive pulmonary blood flow is involved in the pathogenesis of the disease.

Importance of this study:

AV fistula may impose a significant impact on cardiac function and echocardiographic parameters. FIR has been demonstrated to increase access flow of AV fistula in prevalent HD patients. However, its role on newly-created AV fistula is not known. This study will reveal the effect of FIR therapy on echocardiographic parameters, access flow of AVF and endothelial function in patients with end stage renal disease. If FIR therapy is associated with beneficial hemodynamic effect in ESRD patients, it may be considered as a therapeutic modality for improving endothelial function and cardiac performance in ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 18 and 80,
* (2) chronic kidney disease (CKD) stage 5 with clearance of creatinine (CCr) less than 15 ml/min,
* (3) not receiving dialysis or renal transplantation,
* (4) is going to receive creation of AV fistula with the standardized surgical procedures of venous end-to-arterial side anastomosis in the upper extremity.

Exclusion Criteria:

* (1) creation of AV graft or Perm catheter as the type of vascular access,
* (2) heart failure in NYHA Fc III or IV,
* (3) episode of unstable angina, myocardial infarction, cerebrovascular event or receiving percutaneous coronary intervention therapy (PCI; including angioplasty or placement of stent ) within 3 months prior to screening.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Access flow monthly for 3 months and 6th month (0,1st,2nd,3rd and 6th months) and Echocardiographic parameters at 6th month ( 0 and 6th months) | 6 months
  Color Doppler ultrasonography was carried out to measure the access flow of AV fistula with commercially available equipment (Model SSA 340A; Toshiba, Tokyo, Japan). Echocardiographic parameters will be analysed according to the American Society of Echocardiography criteria with a Sonos 5500 sonographic system (Philips, Andover, MA, USA) incorporated with a multi-frequency transducer.Left atrial dimension was determined by M-mode echocardiography.

SECONDARY OUTCOMES:
Plasma asymmetric dimethyl arginine (ADMA) and L-arginine | 6 months (every 3 months)
  Plasma L-arginine and ADMA concentrations were determined by HPLC using precolumn derivatization with o-phthaldialdehyde (OPA) at 0 (before creation of AVF), 3rd and 6th months after creation of AV fistula.

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-CHING LIN, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Lin CC, Yang WC, Chen MC, Liu WS, Yang CY, Lee PC. Effect of far infrared therapy on arteriovenous fistula maturation: an open-label randomized controlled trial. Am J Kidney Dis. 2013 Aug;62(2):304-11. doi: 10.1053/j.ajkd.2013.01.015. Epub 2013 Mar 6. PMID 23474008